CLINICAL TRIAL: NCT03475030
Title: Electronic Medication Adherence Reporting and Feedback During Care Transitions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); TowerView Health (Other)
Responsible Party: Principal Investigator, Jeffrey L. Schnipper, MD.,MPH., Associate Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2016P000241; 1R21HS024587 (AHRQ)
Record Dates: First submitted 2018-03-14; First posted 2018-03-23 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Medication Adherence
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Patients receive usual care and can continue using their existing pharmacy.
- Smart Pillbox (Experimental): Patients receive pre-filled medication trays from Curant Health Pharmacy or the Brigham and Women's Hospital Outpatient Pharmacy. The smart pillbox in which pre-filled medication trays are housed provide automated medication reminders.
  Interventions: Other: pre-filled medication trays; Other: automated medication reminders

INTERVENTIONS:
Other: pre-filled medication trays
  Arms: Smart Pillbox
Other: automated medication reminders
  Arms: Smart Pillbox

SUMMARY:
Patients often have problems with their medications after leaving the hospital and going back home. The goals of this study are to provide a special electronic pill-box with pre-filled weekly medication trays that can alert patients when it is time to take their medications, alert family members (with patients' permission) if there is a problem, and produce a report of medication-taking habits for patients' primary care providers. The investigators will evaluate the effects of this technology on patients' ability to take their medications safely, on the control of chronic conditions like high blood pressure, and also ask patients about any barriers to using this technology in the real world. The investigators hypothesize that a smart pillbox (i) can be successfully implemented in the transitions setting, including engagement of patients, caregivers, and providers in electronically available medication adherence reports; (ii) will decrease medication discrepancies and increase medication adherence in the 6 months after hospital discharge; and (iii) among patients with hypertension, diabetes mellitus, and hyperlipidemia will improve routinely collected measures of disease control.

DETAILED DESCRIPTION:
Adverse drug events are very common after hospitalization and are due to a variety of factors, including misunderstanding of the correct medication regimen and non-adherence with that regimen. The goals of this study are to implement and evaluate a novel "smart pillbox" using health information technology (HIT) to minimize discrepancies in prescribed regimens and improve adherence after hospital discharge. To the investigators' knowledge this type of technology has not been studied in the transitions setting, where there are unique challenges but also tremendous opportunities to engage patients, caregivers, and providers in medication safety and to improve care.

Specific Aims:

1. Implement a smart pillbox intervention for patients discharged from the hospital to the community

   a. Hypothesis 1: a smart pillbox can be successfully implemented in the transitions setting, including engagement of patients, caregivers, and providers in electronically available medication adherence reports
2. Evaluate the effects of the intervention on post-discharge medication discrepancies, medication adherence, and chronic disease management

   1. Hypothesis 2a: a smart pillbox intervention will decrease medication discrepancies and increase medication adherence in the 6 months after hospital discharge
   2. Hypothesis 2b: among patients with hypertension, diabetes mellitus, and hyperlipidemia, a smart pillbox intervention will improve routinely collected measures of disease control
3. Determine barriers and facilitators of implementation of the intervention

To achieve these aims, the investigators will conduct a cluster-randomized controlled trial. This research design will allow for rigorous measurement of medication safety outcomes while minimizing contamination and facilitating education of providers within each practice in the access and use of medication adherence reports created by the smart pillbox and available as a link within the Epic electronic health record (EHR).

This is a Pilot and Feasibility Study focused on several areas, most notably Implementation and Outcomes, although it also evaluates Use (e.g., differences in use and efficacy among in-network providers with access to adherence reports within the EHR and out-of-network providers who do not have access), and Measurement (i.e., a measure of real-time medication adherence that is automatically created by the HIT intervention). The study will generate new knowledge about the benefits of this type of intervention on medication safety and will pave the way for future studies to more precisely quantify the benefits on downstream patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the medicine service of a large, urban hospital
* Taking 5 or more chronic medications

Exclusion Criteria:

* Plan to discharge patient to hospice, rehabilitation, or skilled nursing facility (i.e., not to the community)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Medication Discrepancies | Monthly for the 6 months after discharge
  Number of discrepancies per patient (mean per month)
Medication Adherence | 6 months after discharge
  Proportion of patients with Proportion of Days Covered (PDC) > 80% or Proportion of patients with Daily Polypharmacy Possession Ratio (DPPR) > 80%.

SECONDARY OUTCOMES:
Proportion of regimen in pill trays [intervention arm only] | Biweekly for the 6 months after discharge
  Mean proportion of regimen in pill trays, averaged over all dispense episodes
Biweekly delivery of trays [intervention arm only] | Biweekly for the 6 months after discharge
  Proportion of two-week periods for which delivery was made
Use of adherence reports by patients [intervention arm only] | Cumulative during the 6 months after discharge
  Number of times accessed per patient
Use of adherence reports by caregivers [intervention arm only] | Cumulative during the 6 months after discharge
  Number of times accessed by caregivers, per patient
Use of adherence reports by Partners HealthCare providers [intervention arm only] | Cumulative during the 6 months after discharge
  Number of times accessed by providers, per patient
Actions taken by providers [intervention arm only] | Cumulative during the 6 months after discharge
  Proportion of eligible patients where action taken by providers in response to adherence data when baseline adherence (PDC) is < 80%
Blood Pressure Control (in patients on antihypertensive medications) | Minimum of 6 months
  Last value during 6-month post-discharge study period compared with last value prior to admission. If BP at goal at baseline: maintenance of goal. If BP not at goal at baseline: decrease in systolic and diastolic BP; achievement of goal.
LDL Cholesterol Control (in patients on statins) | Minimum of 6 months
  Last value during 6-month post-discharge study period compared with last value prior to admission. If LDL at goal at baseline: maintenance of goal. If LDL not at goal at baseline: decrease in LDL; achievement of goal.
Diabetes Control (in patients on diabetes medications) | Minimum of 6 months
  Last value during 6-month post-discharge study period compared with last value prior to admission. If A1c at goal at baseline: maintenance of goal. If A1c not at goal at baseline: decrease in A1c; achievement of goal.
14-day adherence [intervention arm only] | 14 day-period
  Proportion of doses opened on schedule from pillbox during any 14-day period

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Schnipper, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shahani A, Nieva HR, Czado K, Shannon E, Gaetani R, Gresham M, Garcia JC, Ganesan H, Cerciello E, Dave J, Jain R, Schnipper JL. An electronic pillbox intervention designed to improve medication safety during care transitions: challenges and lessons learned regarding implementation and evaluation. BMC Health Serv Res. 2022 Oct 30;22(1):1304. doi: 10.1186/s12913-022-08702-y. PMID 36309744